CLINICAL TRIAL: NCT06059170
Title: Rectal Cancer Survivorship: Impact of Low Anterior Resection Syndrome (LARS) on the Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, GIHeelkunde, Clinical nurse specialist digestive oncology, University Hospital, Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/0180
Record Dates: First submitted 2019-05-02; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Rectal Cancer; Low Anterior Resection Syndrome
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Intervention Model Description: cross sectional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QOL, risk factor and therapeutic options (Other): questionnaires
  Interventions: Behavioral: LARS score/ EORTC QLQ C30

INTERVENTIONS:
Behavioral: LARS score/ EORTC QLQ C30 — administering questionnaire

SUMMARY:
Quality of life and risk factors for developing major LARS are explored. Therapeutic options were explored in the cohort experiencing major LARS

DETAILED DESCRIPTION:
Quality of life and risk factors for developing major LARS are explored using the EORTC QLQ C30. Therapeutic options were explored in the cohort experiencing major LARS

ELIGIBILITY:
Inclusion Criteria:

* low anterior resection for rectal cancer between 2006-2016
* Adults

Exclusion Criteria:

* abdomino perineal resection
* patients who do not understand Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment QoL | up to 10 years after rectal resection
  Assessments using questionnaire European Organization for Research and Treatment for Cancer Quality of Life Questionnaire (EORTC QLQ C30)
frequencies of therapeutic options to manage LARS | up to 10 years after rectal resection
  Self developed questionaire to determine what therapeutic options were used to manage LARS
Frequency of LARS | up to 10 years after rectal resection
  Assessment of LARS using validated LARS Score

CONTACTS AND LOCATIONS:
Overall Officials: Piet pattyn, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University hospital Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No
all data are anonymous. only the treating physician has access to the details of the eligible patients